CLINICAL TRIAL: NCT02219802
Title: Revascularization With Paclitaxel-coated Balloon Angioplasty Versus Drug-eluting Stenting in Acute Myocardial Infarction - a Randomized Controlled Trial.
Brief Title: Drug-coated Balloon Versus Drug-eluting Stent in Acute Myocardial Infarction
Acronym: REVELATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Biotronik SE & Co. KG (Industry); Volcano Corporation (Industry)
Responsible Party: Principal Investigator, J.P.R. Herrman, J.P.R.Herrman, MD, PhD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL48495.100.14
Record Dates: First submitted 2014-06-30; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction
Keywords: Coronary artery disease; Acute myocardial infarction; Drug-coated balloon; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-eluting stent (Active Comparator): Treatment of infarct related laesion with a drug-eluting stent
  Interventions: Procedure: Treatment according arm
- Drug-coated balloon (Experimental): After treatment of the infarct related artery with a drug-coated ballon, an additional BMS is advised to be used in case of residual stenosis > 50% or coronary artery dissection type > B.
  Interventions: Procedure: Treatment according arm

INTERVENTIONS:
Procedure: Treatment according arm

SUMMARY:
Rationale: Compared with balloon angioplasty, implantation of bare metal stents (BMS) and drug eluting stents (DES) have shown to reduce repeat target lesion revascularization in primary percutaneous coronary intervention (PPCI). However, this did not result in a reduction of mortality or recurrent myocardial infarction. Furthermore, there are concerns of the occurrence of stent thrombosis. The PAPPA-pilot study, evaluating safety and feasibility of using a drug-coated balloon (DCB) only strategy in PPCI, showed good short- and long-term clinical results, with sustained safety and efficacy at 12 months follow-up. To date little is known about the long-term effects of this treatment modality in STEMI. Besides, angiographic follow-up is of great clinical importance by giving insight on the treated infarct lesion and to assess the functional angioplasty result.

Objective: This randomized controlled, non-inferiority trial is mainly designed to prospectively assess the safety and efficacy of a CE-marked paclitaxel-eluting balloon only strategy vs. third generation DES in the setting of a ST-elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
Rationale: Compared with balloon angioplasty, implantation of bare metal stents (BMS) and drug eluting stents (DES) have shown to reduce repeat target lesion revascularization in primary percutaneous coronary intervention (PPCI). However, this did not result in a reduction of mortality or recurrent myocardial infarction. Furthermore, there are concerns of the occurrence of stent thrombosis. The PAPPA-pilot study, evaluating safety and feasibility of using a drug-coated balloon (DCB) only strategy in PPCI, showed good short- and long-term clinical results, with sustained safety and efficacy at 12 months follow-up. To date little is known about the long-term effects of this treatment modality in STEMI. Besides, angiographic follow-up is of great clinical importance by giving insight on the treated infarct lesion and to assess the functional angioplasty result.

Objective: This randomized controlled, non-inferiority trial is mainly designed to prospectively assess the safety and efficacy of a CE-marked paclitaxel-eluting balloon only strategy vs. third generation DES in the setting of a ST-elevation myocardial infarction (STEMI).

Study design: This is a prospective, single center, non-inferiority, randomized controlled trial.

Study population: All patients presenting with STEMI and suitable for PPCI.

Intervention: PPCI will be performed according to current guidelines. After thrombus aspiration and pre-dilatation, randomization between a DCB only strategy (with bail-out stenting if indicated) and DES will be done by 1:1 ratio. Concomitant medication will be administered according current standards. Control coronary angiography, including measurement of the fractional flow reserve (FFR) of the treated lesion(s), will be performed after 9 months.

Main study parameters/endpoints: The main study parameter is the fractional flow reserve at 9 months follow-up. Secondary study parameters include cardiac death, recurrent myocardial infarction in the target vessel area and ischemia driven target lesion revascularisation at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction eligible for primary PCI:
* > 20 min of chest-pain and at least 1 mm ST-elevation in at least two contiguous leads, a new left bundle branch block or a true posterior myocardial infarction (confirmed by ECG or echocardiography)
* Reperfusion is expected to be feasible within 12 hours after onset of complaints
* Infarct related artery eligible for PPCI and:
* De novo lesion in a native coronary artery
* Reference-vessel diameter ≥ 2.5mm and ≤ 4mm
* Without severe calcification
* Without diameter stenosis of >50% (by visual assessment) after thrombus aspiration and pre-dilatation.

The protocol requires visualization, thrombus aspiration and pre-dilatation of the culprit lesion before inclusion.

Exclusion Criteria:

* Age < 18 years and > 75 years
* History of myocardial infarction
* Known contraindication/resistance for bivalirudin, fondaparinux, heparin, aspirin, prasugrel and/or ticagrelor.
* Participation in another clinical study, interfering with this protocol
* Uncertain neurological outcome e.g. resuscitation
* Intubation/ventilation
* Cardiogenic shock prior to randomization
* Known intracranial disease (mass, aneurysm, AVM, hemorrhagic CVA, ischemic CVA/TIA < 6 months prior to inclusion or ischemic CVA with permanent neurological deficit)
* Gastro-intestinal / urinary tract bleeding < 2 months prior to inclusion
* Refusal to receive blood transfusion
* Planned major surgery within 6 weeks
* Stent implantation < 1 month prior to inclusion
* Expected mortality from any cause within the next 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fractional flow reserve (FFR) | At 9 months follow-up
  Fractional flow reserve is the ratio of mean coronary pressure distal of the treated lesion to mean aortic pressure during maximum hyperemia.

SECONDARY OUTCOMES:
Major adverse cardiac event (MACE) | In-hospital, at 1 and 9 months follow-up and at 2, 3, 4 and 5 year follow-up.
  1. Cardiac death (ARC); defined as any death in which a cardiac cause cannot be excluded.
  2. Recurrent MI in the target vessel area.
  3. Ischemia driven target lesion revascularization (PCI within 5 mm of the treated segment in case of balloon, or stent area borders in case of stent, or CABG of the target vessel).
Angiographic endpoint: iFR | At 9 months follow-up.
ST-segment resolution | 90 minutes after initial procedure
  ST-segment resolution post-initial procedure at 90 minutes, defined as the ST-segment deviation resolution in only the single lead showing maximum deviation.
Non-coronary artery bypass grafting major bleeding | At 1 month follow-up
  * Intracranial, intraocular, intra-articular or retroperitoneal bleeding
  * Access site bleed requiring intervention/surgery
  * Hematoma ≥ 5 cm
  * Hemoglobin (Hgb) ≥4 g/dL without an overt source
  * Hgb ≥3 g/dL with an overt source
  * Operation for bleeding
  * Any blood transfusions
Stent thrombosis | During follow-up
  * Definite or confirmed stent thrombosis: Angiographic confirmation of vessel occlusion or thrombus formation within, or adjacent to, the stented segment or proven stent thrombosis at autopsy.
  * Probable stent thrombosis: Unexplained death within 30 days or target vessel recurrent MI without angiographic confirmation.
  * Possible stent thrombosis: Unexplained death after 30 days.
Angiographic endpoint: TIMI flow | At 9 months follow-up
Angiographic endpoint: late lumen loss | At 9 months follow-up
Angiographic endpoint: minimal lumen diameter | At 9 months follow-up
Angiographic endpoint: diameter stenosis | At 9 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: R. J. van der Schaaf, MD, PhD, Principal Investigator — OLVG
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Zijlstra F, Hoorntje JC, de Boer MJ, Reiffers S, Miedema K, Ottervanger JP, van 't Hof AW, Suryapranata H. Long-term benefit of primary angioplasty as compared with thrombolytic therapy for acute myocardial infarction. N Engl J Med. 1999 Nov 4;341(19):1413-9. doi: 10.1056/NEJM199911043411901. PMID 10547403
- [Background] Stone GW, Grines CL, Browne KF, Marco J, Rothbaum D, O'Keefe J, Hartzler GO, Overlie P, Donohue B, Chelliah N, et al. Predictors of in-hospital and 6-month outcome after acute myocardial infarction in the reperfusion era: the Primary Angioplasty in Myocardial Infarction (PAMI) trail. J Am Coll Cardiol. 1995 Feb;25(2):370-7. doi: 10.1016/0735-1097(94)00367-y. PMID 7829790
- [Background] Zijlstra F, de Boer MJ, Hoorntje JC, Reiffers S, Reiber JH, Suryapranata H. A comparison of immediate coronary angioplasty with intravenous streptokinase in acute myocardial infarction. N Engl J Med. 1993 Mar 11;328(10):680-4. doi: 10.1056/NEJM199303113281002. PMID 8433726
- [Background] Mintz GS. Remodeling and Restenosis: Observations from Serial Intravascular Ultrasound Studies. Curr Interv Cardiol Rep. 2000 Nov;2(4):316-325. PMID 11096682
- [Background] Zhu MM, Feit A, Chadow H, Alam M, Kwan T, Clark LT. Primary stent implantation compared with primary balloon angioplasty for acute myocardial infarction: a meta-analysis of randomized clinical trials. Am J Cardiol. 2001 Aug 1;88(3):297-301. doi: 10.1016/s0002-9149(01)01645-9. No abstract available. PMID 11472712
- [Background] De Luca G, Suryapranata H, Stone GW, Antoniucci D, Biondi-Zoccai G, Kastrati A, Chiariello M, Marino P. Coronary stenting versus balloon angioplasty for acute myocardial infarction: a meta-regression analysis of randomized trials. Int J Cardiol. 2008 May 7;126(1):37-44. doi: 10.1016/j.ijcard.2007.03.112. Epub 2007 Jun 4. PMID 17544528
- [Background] Suryapranata H, De Luca G, van 't Hof AW, Ottervanger JP, Hoorntje JC, Dambrink JH, Gosselink AT, Zijlstra F, de Boer MJ. Is routine stenting for acute myocardial infarction superior to balloon angioplasty? A randomised comparison in a large cohort of unselected patients. Heart. 2005 May;91(5):641-5. doi: 10.1136/hrt.2004.056705. PMID 15831652
- [Background] Laarman GJ, Suttorp MJ, Dirksen MT, van Heerebeek L, Kiemeneij F, Slagboom T, van der Wieken LR, Tijssen JG, Rensing BJ, Patterson M. Paclitaxel-eluting versus uncoated stents in primary percutaneous coronary intervention. N Engl J Med. 2006 Sep 14;355(11):1105-13. doi: 10.1056/NEJMoa062598. PMID 16971717
- [Background] Kastrati A, Dibra A, Spaulding C, Laarman GJ, Menichelli M, Valgimigli M, Di Lorenzo E, Kaiser C, Tierala I, Mehilli J, Seyfarth M, Varenne O, Dirksen MT, Percoco G, Varricchio A, Pittl U, Syvanne M, Suttorp MJ, Violini R, Schomig A. Meta-analysis of randomized trials on drug-eluting stents vs. bare-metal stents in patients with acute myocardial infarction. Eur Heart J. 2007 Nov;28(22):2706-13. doi: 10.1093/eurheartj/ehm402. Epub 2007 Sep 27. PMID 17901079
- [Background] De Luca G, Stone GW, Suryapranata H, Laarman GJ, Menichelli M, Kaiser C, Valgimigli M, Di Lorenzo E, Dirksen MT, Spaulding C, Pittl U, Violini R, Percoco G, Marino P. Efficacy and safety of drug-eluting stents in ST-segment elevation myocardial infarction: a meta-analysis of randomized trials. Int J Cardiol. 2009 Apr 3;133(2):213-22. doi: 10.1016/j.ijcard.2007.12.040. Epub 2008 Apr 3. PMID 18394731
- [Background] Degertekin M, Serruys PW, Tanabe K, Lee CH, Sousa JE, Colombo A, Morice MC, Ligthart JM, de Feyter PJ. Long-term follow-up of incomplete stent apposition in patients who received sirolimus-eluting stent for de novo coronary lesions: an intravascular ultrasound analysis. Circulation. 2003 Dec 2;108(22):2747-50. doi: 10.1161/01.CIR.0000103666.25660.77. Epub 2003 Nov 24. PMID 14638542
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Nakazawa G, Finn AV, Joner M, Ladich E, Kutys R, Mont EK, Gold HK, Burke AP, Kolodgie FD, Virmani R. Delayed arterial healing and increased late stent thrombosis at culprit sites after drug-eluting stent placement for acute myocardial infarction patients: an autopsy study. Circulation. 2008 Sep 9;118(11):1138-45. doi: 10.1161/CIRCULATIONAHA.107.762047. Epub 2008 Aug 25. PMID 18725485
- [Background] Vink MA, Dirksen MT, Suttorp MJ, Tijssen JG, van Etten J, Patterson MS, Slagboom T, Kiemeneij F, Laarman GJ. 5-year follow-up after primary percutaneous coronary intervention with a paclitaxel-eluting stent versus a bare-metal stent in acute ST-segment elevation myocardial infarction: a follow-up study of the PASSION (Paclitaxel-Eluting Versus Conventional Stent in Myocardial Infarction with ST-Segment Elevation) trial. JACC Cardiovasc Interv. 2011 Jan;4(1):24-9. doi: 10.1016/j.jcin.2010.11.003. PMID 21251625
- [Background] Hong MK, Mintz GS, Lee CW, Kim YH, Lee SW, Song JM, Han KH, Kang DH, Song JK, Kim JJ, Park SW, Park SJ. Incidence, mechanism, predictors, and long-term prognosis of late stent malapposition after bare-metal stent implantation. Circulation. 2004 Feb 24;109(7):881-6. doi: 10.1161/01.CIR.0000116751.88818.10. Epub 2004 Feb 16. PMID 14967732
- [Background] Gonzalo N, Barlis P, Serruys PW, Garcia-Garcia HM, Onuma Y, Ligthart J, Regar E. Incomplete stent apposition and delayed tissue coverage are more frequent in drug-eluting stents implanted during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction than in drug-eluting stents implanted for stable/unstable angina: insights from optical coherence tomography. JACC Cardiovasc Interv. 2009 May;2(5):445-52. doi: 10.1016/j.jcin.2009.01.012. PMID 19463469
- [Background] Herdeg C, Oberhoff M, Baumbach A, Blattner A, Axel DI, Schroder S, Heinle H, Karsch KR. Local paclitaxel delivery for the prevention of restenosis: biological effects and efficacy in vivo. J Am Coll Cardiol. 2000 Jun;35(7):1969-76. doi: 10.1016/s0735-1097(00)00614-8. PMID 10841250
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Two year follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2008 Oct;97(10):773-81. doi: 10.1007/s00392-008-0682-5. Epub 2008 Jun 5. PMID 18536865
- [Background] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- [Background] De Labriolle A, Pakala R, Bonello L, Lemesle G, Scheinowitz M, Waksman R. Paclitaxel-eluting balloon: from bench to bed. Catheter Cardiovasc Interv. 2009 Apr 1;73(5):643-52. doi: 10.1002/ccd.21895. PMID 19309715
- [Background] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2010 Mar;99(3):165-74. doi: 10.1007/s00392-009-0101-6. Epub 2010 Jan 6. PMID 20052480
- [Background] Vos NS, Dirksen MT, Vink MA, van Nooijen FC, Amoroso G, Herrman JP, Kiemeneij F, Patterson MS, Slagboom T, van der Schaaf RJ. Safety and feasibility of a PAclitaxel-eluting balloon angioplasty in Primary Percutaneous coronary intervention in Amsterdam (PAPPA): one-year clinical outcome of a pilot study. EuroIntervention. 2014 Sep;10(5):584-90. doi: 10.4244/EIJV10I5A101. PMID 25256200
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] De Bruyne B, Pijls NH, Bartunek J, Kulecki K, Bech JW, De Winter H, Van Crombrugge P, Heyndrickx GR, Wijns W. Fractional flow reserve in patients with prior myocardial infarction. Circulation. 2001 Jul 10;104(2):157-62. doi: 10.1161/01.cir.104.2.157. PMID 11447079
- [Background] Bech GJ, De Bruyne B, Pijls NH, de Muinck ED, Hoorntje JC, Escaned J, Stella PR, Boersma E, Bartunek J, Koolen JJ, Wijns W. Fractional flow reserve to determine the appropriateness of angioplasty in moderate coronary stenosis: a randomized trial. Circulation. 2001 Jun 19;103(24):2928-34. doi: 10.1161/01.cir.103.24.2928. PMID 11413082
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Legrand V, Mancini GB, Bates ER, Hodgson JM, Gross MD, Vogel RA. Comparative study of coronary flow reserve, coronary anatomy and results of radionuclide exercise tests in patients with coronary artery disease. J Am Coll Cardiol. 1986 Nov;8(5):1022-32. doi: 10.1016/s0735-1097(86)80377-1. PMID 3760377
- [Background] Zijlstra F, Fioretti P, Reiber JH, Serruys PW. Which cineangiographically assessed anatomic variable correlates best with functional measurements of stenosis severity? A comparison of quantitative analysis of the coronary cineangiogram with measured coronary flow reserve and exercise/redistribution thallium-201 scintigraphy. J Am Coll Cardiol. 1988 Sep;12(3):686-91. doi: 10.1016/s0735-1097(88)80057-3. PMID 3403826
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] Nam CW, Hur SH, Cho YK, Park HS, Yoon HJ, Kim H, Chung IS, Kim YN, Kim KB, Doh JH, Koo BK, Tahk SJ, Fearon WF. Relation of fractional flow reserve after drug-eluting stent implantation to one-year outcomes. Am J Cardiol. 2011 Jun 15;107(12):1763-7. doi: 10.1016/j.amjcard.2011.02.329. Epub 2011 Apr 8. PMID 21481828
- [Background] Klauss V, Erdin P, Rieber J, Leibig M, Stempfle HU, Konig A, Baylacher M, Theisen K, Haufe MC, Sroczynski G, Schiele T, Siebert U. Fractional flow reserve for the prediction of cardiac events after coronary stent implantation: results of a multivariate analysis. Heart. 2005 Feb;91(2):203-6. doi: 10.1136/hrt.2003.027797. PMID 15657233
- [Background] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731
- [Background] Jeremias A, Maehara A, Genereux P, Asrress KN, Berry C, De Bruyne B, Davies JE, Escaned J, Fearon WF, Gould KL, Johnson NP, Kirtane AJ, Koo BK, Marques KM, Nijjer S, Oldroyd KG, Petraco R, Piek JJ, Pijls NH, Redwood S, Siebes M, Spaan JAE, van 't Veer M, Mintz GS, Stone GW. Multicenter core laboratory comparison of the instantaneous wave-free ratio and resting Pd/Pa with fractional flow reserve: the RESOLVE study. J Am Coll Cardiol. 2014 Apr 8;63(13):1253-1261. doi: 10.1016/j.jacc.2013.09.060. Epub 2013 Nov 6. PMID 24211503
- [Background] Mehran R, Lansky AJ, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Wong SC, Nikolsky E, Gambone L, Vandertie L, Parise H, Dangas GD, Stone GW; HORIZONS-AMI Trial Investigators. Bivalirudin in patients undergoing primary angioplasty for acute myocardial infarction (HORIZONS-AMI): 1-year results of a randomised controlled trial. Lancet. 2009 Oct 3;374(9696):1149-59. doi: 10.1016/S0140-6736(09)61484-7. Epub 2009 Aug 28. PMID 19717185
- [Background] Cortese B, Picchi A, Micheli A, Ebert AG, Parri F, Severi S, Limbruno U. Comparison of prolonged bivalirudin infusion versus intraprocedural in preventing myocardial damage after percutaneous coronary intervention in patients with angina pectoris. Am J Cardiol. 2009 Oct 15;104(8):1063-8. doi: 10.1016/j.amjcard.2009.06.005. PMID 19801025
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Derived] Vos NS, Fagel ND, Amoroso G, Herrman JR, Patterson MS, Piers LH, van der Schaaf RJ, Slagboom T, Vink MA. Paclitaxel-Coated Balloon Angioplasty Versus Drug-Eluting Stent in Acute Myocardial Infarction: The REVELATION Randomized Trial. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1691-1699. doi: 10.1016/j.jcin.2019.04.016. Epub 2019 May 21. PMID 31126887